CLINICAL TRIAL: NCT06773039
Title: Assessment of Toxicity and Outcomes of Different Therapeutic Strategies in Patients With Head and Neck Neoplasms Treated With Radiotherapy at the IRCCS Azienda Ospedaliero-Universitaria di Bologna
Brief Title: Assessment of Different Therapeutic Strategies in Patients With Head and Neck Neoplasms Treated With Radiotherapy
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: PORTO
Record Dates: First submitted 2024-12-01; First posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2024-10

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a monocentric observational study aimed at collecting data related to the radiotherapy treatment of head and neck neoplasms. The purpose of the study is to systematically gather data on radiotherapy for head and neck neoplasms to evaluate tumor response and potential toxicity in relation to dosages and techniques used, the combination with other therapies, disease characteristics, and the psychological impact of the proposed treatments.

Additionally, collecting data on both disease characteristics and pre-existing conditions in a large sample may allow for the assessment of any correlation with radiation-induced toxicities, with the goal of predicting and preventing them in a personalized manner in the future.

The study's aim is thus to evaluate tumor response and any potential toxicity following radiotherapy treatment concerning treatment modalities, dosages, and techniques used, for both new diagnoses and cases already diagnosed and treated since January 1, 2000, at the Radiotherapy Unit of the S. Orsola-Malpighi Polyclinic. The structured data collection necessary for evaluating the objectives will cover the observation period from January 1, 2000, to December 15, 2030, involving approximately 3,000 patients. Participation in the study solely involves the structured collection of certain information already present in your medical records, as well as data related to clinical exams, radiological imaging, and therapies, without any modifications to standard clinical practice. Participation in the study incurs no costs and will not be compensated in any way. There are no risks or inconveniences associated with participating in this study. Enrolled patients will not receive any direct benefit from this study, as it is purely a data collection effort. The collected data will enhance understanding of the factors associated with treatment outcomes, ultimately leading to improved management of each individual patient.

DETAILED DESCRIPTION:
Head and neck tumors refer to neoplasms that originate in the nasal cavities and paranasal sinuses, rhinopharynx/oropharynx/hypopharynx, salivary glands, oral cavity, and larynx, mostly represented by squamous cell carcinomas. Head and neck tumors account for 4.9% of all malignant tumors worldwide.

Treatment is mostly multimodal; the main therapeutic options include surgery, systemic therapy, and radiotherapy. Various treatments may serve as primary or adjuvant therapy depending on the specific neoplasm and the strategy adopted.

Regarding radiotherapy, it is often used in combination with other treatments depending on the stage, location of the disease, risk factors, or in a palliative setting. Dosages, fractionation, and techniques vary based on the type of neoplasm being treated and the purpose of the therapy (adjuvant, radical, palliative), as do the possible acute and late toxicities related to the treatment characteristics.

The purpose of the study is to systematically collect data related to radiotherapy treatment in head and neck neoplasms in order to evaluate outcomes in relation to dosages, fractionation, and techniques used, as well as combinations with other therapies and disease characteristics. Additionally, collecting data on both disease characteristics and treatments in a large sample may enable the assessment of any potential correlation with radiation-induced toxicities, allowing for future prediction and personalized prevention.

Enrolled patients will not have any direct benefit or harm from their participation in the study, as it is solely a data collection effort. Conversely, these data may lead to new insights that improve the management of the analyzed neoplastic diseases in the future.

The study thus aims to evaluate outcomes, toxicity, and the psychological impact on patients related to radiotherapy treatment concerning treatment settings, dosages, and techniques used, for both new diagnoses and cases already diagnosed and treated since January 1, 2000, at the Radiotherapy Unit of the S. Orsola Polyclinic. The structured data collection necessary for evaluating the objectives will cover the observation period from January 1, 2000, to December 15, 2030, involving approximately 3,000 patients (2,000 for the retrospective phase and 1,000 for the prospective phase).

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes, aged ≥ 18 years, with new or previous diagnosis of malignant neoplasm of the head and neck, from January 1, 2000, treated at the Radiotherapy Unit of the S. Orsola Polyclinic
* Obtaining informed consent

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with new or previous diagnosis of malignant neoplasm of the head and neck
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2021-10-28 (Actual); Primary Completion 2030-11-15 (Estimated); Study Completion 2030-12-15 (Estimated)

PRIMARY OUTCOMES:
Evaluate the correlation of therapy response | From enrollment to the last follow-up at 12 months
  Evaluate the correlation of therapy response with other parameters in the radiotherapy treatment of head and neck neoplasms, considering the treatment setting, dosages, and techniques used

SECONDARY OUTCOMES:
Acute toxicity | immediate to 6 months after radiotherapy
  acute toxicity after radiotherapy, evaluated according to CTCAE v.5
Late toxicity | from 6 months after radiotherapy, through study completion, an average of 1 year
  late toxicity after completion of treatments, evaluated according to CTCAE v.5
Impact on the patient's quality of life | From enrollment to the last follow-up at 12 months
  The impact on patients' quality of life will be assessed through the submission of questionnaires (FACT H&N)
Retreatments | During the follow-ups, up to the last one at 12 months
  Retreatments yes or not
Disease-free survival | During the follow-ups, up to the last one at 12 months
  Disease-free survival assessed based on the presence or absence of local, nodal, or metastatic recurrences
Overall survival | From enrollment to the last follow-up at 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Alessio Giuseppe Morganti, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero - Universitaria di Bologna, Bologna, Italy